CLINICAL TRIAL: NCT00955643
Title: Periodontal Therapy in Severe Cases of Periodontitis: Preliminary Findings of Non-surgical Instrumentation With or Without Hyperbaric Oxygen Therapy (HBOT)
Brief Title: Periodontal Treatment Associated With Hyperbaric Oxygen Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Bahiana de Medicina e Saude Publica (Other)
Responsible Party: EBMSP, Bahiana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HBOT900208-06
Record Dates: First submitted 2009-08-07; First posted 2009-08-10 (Estimated); Last update posted 2009-08-10 (Estimated); Status verified 2009-08

CONDITIONS: Periodontal Disease
Keywords: periodontitis; hyperbaric oxygen therapy
MeSH Terms: conditions — Periodontal Diseases; Periodontitis | interventions — Oxygen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- hyperbaric therapy (Experimental): Hyperbaric therapy by oxygen
  Interventions: Other: oxygen
- dental scaling and root planing (Experimental): dental scaling and cleaning
  Interventions: Other: other

INTERVENTIONS:
Other: oxygen
  Arms: hyperbaric therapy
Other: other
  Arms: dental scaling and root planing

SUMMARY:
Evaluation of the clinical effect of hyperbaric oxygen therapy (HBOT) adjunctively to scaling and root planing (SRP) in the treatment of severe case of chronic periodontitis.

DETAILED DESCRIPTION:
Materials and Methods: In 20 patients diagnosed with severe generalized chronic periodontitis (pockets>7mm) with bleeding on probing, SRP was rendered in all pockets. Additionally, five consecutive hyperbaric sessions were administered in 10 patients after random allocation (SRP+HBOT). Clinical parameters were assessed at baseline up to 6 months: plaque index (PI), bleeding on probing, probing depth, clinical attachment level and BANA test.

Results: SRP+HBOT resulted in greater probing reduction and attachment gain than SRP alone 3 months after treatment (p<0.001). The BANA test was negative after 1 week only for sites in the SRP+HBOT group (p<0.05). However SRP+HBOT failed to show a significant difference from SRP group after 3 months were all BANA sites became negative (p>0.05).

Conclusion: These preliminary data suggest that hyperbaric oxygen therapy had a short-term beneficial effect on pocket reduction and bacterial elimination, and may be considered a potential therapy option to improve the clinical outcomes of scaling in severe cases of chronic periodontitis.

ELIGIBILITY:
Inclusion criteria:

* This preliminary (pilot) study was designed with twenty subjects (12 men, 8 women, mean age 37.3 years) selected from a pool of 360 patients referred to the Periodontal Clinic of the School of Dentistry at Bahian Science Foundation (FBDC, Bahia, Brazil).
* The patients had an initial diagnosis of severe generalized chronic periodontitis (AAP 1999).

Exclusion criteria:

* Patients were excluded according to the following criteria:

  * smoking
  * pregnancy or lactation
  * antibiotics or periodontal treatment within the last 6 months
  * a diagnosis of aggressive periodontitis
  * trauma from occlusion or endodontic lesions
* According to an accurate clinical examination performed by a hyperbaric medical doctor (MD), the HBOT contra-indications (Iazzeti & Mantovani 1998) served as exclusion criteria.
* The only absolute contraindication to hyperbaric oxygen therapy was from patients with untreated pneumothorax
* Relative contraindications were considered:

  * upper respiratory infections
  * high fevers
  * emphysema with CO2 retention
  * historic of thoracic surgery
  * malignant disease and middle ear barotrauma
* Patients taking or have recently taken the following drugs:

  * doxorubicin (Adriamycin®)
  * disulfiram (Antabuse®)
  * Cis-platinum and mafenide acetate (Sulfamylon®).

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2002-03; Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- EBMSP Central Clinic, Salvador, Estado de Bahia, Brazil